CLINICAL TRIAL: NCT03201224
Title: Image Transmission Applied to Organ Transplant: Before-after Study of the Device of the Effectiveness
Brief Title: Image Transmission Applied to Organ Transplant: Before-after Study of the Effectiveness of the Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PREPS - Cristal Images
Record Dates: First submitted 2017-06-13; First posted 2017-06-28 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2018-09

CONDITIONS: Transplantation, Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group without image transmission: "Before" Group
- Group with image transmission: "After" Group
  Interventions: Device: "After" Group

INTERVENTIONS:
Device: "After" Group
  Groups: Group with image transmission

SUMMARY:
In the complex process of organ transplant, two of the major steps are:

1. evaluation of the organs of potential donors in health institutions:
2. proposing grafts to the transplant teams, according to rules defined at the national level.

In the absence of the possibility of transmitting the images between the deceased donor sites and the transplant teams, the visualization of these examinations does not take part in the decision-making of the transplant team. This leads in the displacement of the transplant team in order to verify the grafts after acceptance of the graft proposal.

The "Cristal Image" project is a visualisation project for the transplant teams, in real time, at the time of the proposal of the graft so that they can give an opinion (acceptance, refusal) in less than 20 minutes (legal delay for a vital organ) after analyzing the medical records provided and the imaging data (scanner, ultrasound (s), coronary angiography, etc.).

The hypothesis of the project is that the implementation of a secure image transmission (complete anonymisation of the data of the donor) before the acceptance by the team, will allow an optimization of the use of the qualified organs by reducing risks, unnecessary displacement of transplant surgical teams, and securing the allocation of organs to recipient patients.

ELIGIBILITY:
Inclusion Criteria:

* French Donors who died in brain death, at least one organ of which was proposed for transplantation (kidneys, liver, heart, lung); Recipients transplanted during the same periods.

Exclusion Criteria:

* Donors who died after cardiac arrest
* Donors taken care in a foreign country or outside the Metropolitan France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All health institutions authorized for organ transplantation in metropolitan France are concerned.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of successful organ transplantation among those sampled. | 3 months after transplantation for kidney, 1 year after transplantation for the other organs

SECONDARY OUTCOMES:
Number of assigned organs but not sampled | Immediately after the decision of the transplant team
Number of useless graft transportation | Immediately after the decision of the transplant team
Number of useless graft team transportation | Immediately after the decision of the transplant team
Mortality or function stop | 1 year after transplantation
Duration of the graft assignment | Immediately after graft assignment
Cost of sampling process | Immediately after the sampling process
Use of image transmission by the graft team | Immediately after decision of the transplant team to accept or not the graft

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris - DRCD URC Eco
Locations (1):
- Agence de la biomédecine, Saint-Denis, France

REFERENCES:
- [Background] Reddy MS, Bhati C, Neil D, Mirza DF, Manas DM. National Organ Retrieval Imaging System: results of the pilot study. Transpl Int. 2008 Nov;21(11):1036-44. doi: 10.1111/j.1432-2277.2008.00720.x. PMID 18764835
- [Background] Rosenkrantz AB, Campbell N, Wehrli N, Triolo MJ, Kim S. New OPTN/UNOS classification system for nodules in cirrhotic livers detected with MR imaging: effect on hepatocellular carcinoma detection and transplantation allocation. Radiology. 2015 Feb;274(2):426-33. doi: 10.1148/radiol.14140069. Epub 2014 Oct 7. PMID 25299785
- [Background] Furlow B. Solid organ donation and transplantation. Radiol Technol. 2012 Mar-Apr;83(4):371-89. PMID 22461345
- [Background] Fregeville A, De Bazelaire C, Zagdanski A, Albiter M, Desgrandchamps F, De Kerviler E. [Value of whole body CTA in the management of brain-dead patients]. J Radiol. 2010 Jan;91(1 Pt 1):37-44. doi: 10.1016/s0221-0363(10)70004-4. French. PMID 20212375
- [Background] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558
- [Derived] Zarca K, Dupont JK, Jacoud L, Bulsei J, Huot O, Logerot H, Durand-Zaleski I. Effectiveness and efficiency of teleimaging in the transplantation process: a mixed method protocol. BMC Health Serv Res. 2019 Sep 18;19(1):672. doi: 10.1186/s12913-019-4488-0. PMID 31533713